CLINICAL TRIAL: NCT04016064
Title: Evaluation of Temperature and Healing in Treatment of Gingival Enlargement Using Different Gingivectomy Techniques
Brief Title: Temperature and Healing in Treatment of Gingival Enlargement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, mehmet murat taskan, Assistant Professor, Tokat Gaziosmanpasa University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: OMU KAEK 2012/167
Record Dates: First submitted 2019-07-08; First posted 2019-07-11 (Actual); Last update posted 2019-07-11 (Actual); Status verified 2019-07

CONDITIONS: Gingival Enlargement
Keywords: gingival enlargement, Er:YAG, Nd:YAG, electrosurgery
MeSH Terms: conditions — Gingival Hyperplasia; Hyperthermia | interventions — Lasers, Solid-State

STUDY DESIGN:
Intervention Model Description: The present study was designed as a controlled clinical study with a randomized design. The study protocol was approved by the local ethical committee of Clinical Studies of Ondokuz Mayis University. The study population consisted of 37 participants (19 women, age 23.10±2.78, 18 men age 21.11±2.63).
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1; (Other): Er:YAG laser
  Interventions: Procedure: Er:YAG LASER, Nd:YAG laser, elctrosurgery, conventional surgery
- group 2 (Other): Nd:YAG laser
  Interventions: Procedure: Er:YAG LASER, Nd:YAG laser, elctrosurgery, conventional surgery
- group 3 (Other): Electrosurgery
  Interventions: Procedure: Er:YAG LASER, Nd:YAG laser, elctrosurgery, conventional surgery

INTERVENTIONS:
Procedure: Er:YAG LASER, Nd:YAG laser, elctrosurgery, conventional surgery — 1. Er: YAG laser (Fotana AT Fidelis III, Ljubljana, Slovenia) 200 mj, 10 Hz, 2 Watt and VLP (long pulse, 1000 μs); 1.3 mm diameter, 8 mm long cylindrical, a sapphire tip was used with air cooling and water irrigation.
  2. Nd: YAG laser (Fotana AT Fidelis III, Ljubljana, Slovenia) was applied at 4 watts, 50 Hz, 300 μm microfiber tip and SP (short pulse: 180 μs) settings.
  3. Electrosurgical (Servotome Classic System, High Frequency Surgical Equipment, Satelec, France).
  4. Conventional surgical method was applied with hand instruments and gingivectomy knives.

SUMMARY:
Aim: Gingival enlargement is a common clinical condition which requires surgical approaches to alleviating these enlargement areas. The aim of this study was to investigate epithelization, gingival temperature, inflammation and pain levels in post-operative healing process in 4 different gingivectomy techniques including Er:YAG laser, Nd:YAG laser, electrosurgery and conventional gingivectomy in treatment of chronic inflammatory gingival enlargements.

Material and Method: A split-mouth designed study was conducted on 37 systemically healthy patients consisting of 19 females and 18 males, who had gingival enlargement areas on the left and right of maxillary and mandibular anterior regions. Gingival crevicular fluid (GCF) samples were collected, clinical periodontal parameters and gingival temperature levels were recorded at baseline and in the postoperative period. The gingival temperature was measured during surgical procedures. Gingival temperature and epithelization levels in 3rd, 7th, 10th and 15th days; GCF levels in 15th, 30th, and 90th days and pain levels in 2nd and 8th hours and between 1st-7th days of post-operative healing process were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* systemically healthy individuals
* the existence of at least 20 functioning teeth, the existence of chronic inflammatory gingival enlargement in anterior quadrants.

Exclusion Criteria:

* pregnancy/lactation
* drug use, previous periodontal therapy within 6 months
* previous antibiotic use within 6 months, smoking
* the existence of attachment/bone loss. .

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2013-05-01 (Actual); Study Completion 2013-12-01 (Actual)

PRIMARY OUTCOMES:
Epithelization | Epithelization was evaluated at postoperative 7th day
  Wound surface epithelization in the healing process was evaluated with a staining solution (Mira-2-tone, GMBH & Co., Duisburg, Germany). (O. Ozcelik et al., 2008)

SECONDARY OUTCOMES:
Gingival temperature | The gingival temperature was measured during surgical procedures
  The temperature measurement during the process was performed by an infrared thermometer (Optris GMBH, Manuel LS, Berlin, Germany). The device had a measurement and recording range from -35 ° C to 900 ° C, optical resolution 75: 1, thermal resolution 0.1 ° C, waveband range 8-14, USB interface and graphical software program.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No